CLINICAL TRIAL: NCT01876615
Title: A Randomized, Open-Label, Single-dosing and Cross-over Clinical Trial to Investigate the Safety and Pharmacokinetic Drug-Drug Interaction of YH4808 and Diclofenac in Healthy Male Volunteers
Brief Title: Pharmacokinetic Drug Interaction Between YH4808 and Diclofenac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: YH4808-109
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: safety/tolerability and pharmacokinetics/pharmacodynamics
MeSH Terms: interventions — YH4808; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- YH4808 or Diclofenac or YH4808+Diclofenac(arm 1) (Experimental): 6 arm, 3 Sequence design
  * YH4808 or Diclofenac or YH4808+Diclofenac
  * 3 week wash out period is between each period.
  Interventions: Drug: YH4808; Drug: Diclofenac; Drug: YH4808+Diclofenac
- YH4808 or Diclofenac or YH4808+Diclofenac (arm 2) (Experimental): 6 arm, 3 Sequence design
  * YH4808 or Diclofenac or YH4808+Diclofenac
  * 3 week wash out period is between each period.
  Interventions: Drug: YH4808; Drug: Diclofenac; Drug: YH4808+Diclofenac
- YH4808 or Diclofenac or YH4808+Diclofenac (arm 3) (Experimental): 6 arm, 3 Sequence design
  * YH4808 or Diclofenac or YH4808+Diclofenac
  * 3 week wash out period is between each period.
  Interventions: Drug: YH4808; Drug: Diclofenac; Drug: YH4808+Diclofenac
- YH4808 or Diclofenac or YH4808+Diclofenac (arm 4) (Experimental): 6 arm, 3 Sequence design
  * YH4808 or Diclofenac or YH4808+Diclofenac
  * 3 week wash out period is between each period.
  Interventions: Drug: YH4808; Drug: Diclofenac; Drug: YH4808+Diclofenac
- YH4808 or Diclofenac or YH4808+Diclofenac (arm5) (Experimental): 6 arm, 3 Sequence design
  * YH4808 or Diclofenac or YH4808+Diclofenac
  * 3 week wash out period is between each period.
  Interventions: Drug: YH4808; Drug: Diclofenac; Drug: YH4808+Diclofenac
- YH4808 or Diclofenac or YH4808+Diclofenac (arm6) (Experimental): 6 arm, 3 Sequence design
  * YH4808 or Diclofenac or YH4808+Diclofenac
  * 3 week wash out period is between each period.
  Interventions: Drug: YH4808; Drug: Diclofenac; Drug: YH4808+Diclofenac

INTERVENTIONS:
Drug: YH4808 — experimental drug
Drug: Diclofenac — Depain tablet 25mg
  Other Names: Depain tablet 25mg
Drug: YH4808+Diclofenac

SUMMARY:
The objective of this study is to compare pharmacokinetics after single oral administration of YH4808 and Diclofenac each separately versus coadministration of YH4808 and Diclofenac in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* healthy male age 20 to 45 over 55kg with Ideal body weight(IBW)
* No clinically important abnormal physical findings at the screening examination
* Subject who has no congential, chronic disease and disease symptoms in medical examination result
* Subject who is judged to be eligible by principal inverstigator or sub-investigator according to various reasons includiong ther abnorminal test results(clinical laboratory test, 12-lead GCG etc)
* Ability to communicate well with the inverstigator and to comply with the requremetns of the entire study
* Willingness to give written informed consent(prior to any study-related procedures beinging performed) and to be able to adhere to the study restrictions and examination schedule

Exclusion Criteria:

* Suject who has history or presence of clinically significant diseases in liver, kidney, gastrointestinal tract, nervous system, respiratory system, endocrine system, blood tumor, cardiovascular, urinary system, and mental disorder
* Subject who is hypersensitive to components contained in YH4808 or declofenac or related drug(ex. rebamipide, revaprazan, NSID etc)
* Medical history of gastrointestinal disease or acid restraining surgery, gastric/ esophagus surgery(excluding appendectomy, hernia surgery)
* Subject who has history of drug dependence or using that drug
* Subject who had taken usual dose of any prescription durgs within 14 days before the treatment or who had used usual dose of OTC drugs within 7 days before the treatment
* Subject who participated in antoher clinical trial within 2 monthes before enrolling in this study
* subject who donated whole blood within 2 months or component blood within 1 month before the treatment
* Subject who drank over 21unit/week(1 unit= 10g of alcohol) or were not able to refrain from drinking alcohol during study days
* Subject who stopped smoking within 3 months before the treatment or detected cotinine in urine test
* Subject with clinically significant observations considered as unsuitable based on medical judgment by the investigators

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cmax of YH4808 | 18 points up to Day 2 or Day 3
AUClast of YH4808 | 18 points up to Day 3

SECONDARY OUTCOMES:
AUCinf of YH4808 | 18 points up to Day 3
AUCinf of Diclofenac | 16points up to Day 2
t1/2 of YH4808 | 18 points up to Day 3
t1/2 of Diclofenac | 16 points up to Day 2
Tmax of YH4808 | 18 points up to Day 3
Tmax of Diclofenac | 16 points up to Day 2
Metabolic ratio | 18 points up to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Janghee Hong, Professor, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea